CLINICAL TRIAL: NCT06081361
Title: A Multicenter, Randomized, Open-Label Study To Evaluate The Efficacy And Safety Of A Contezolid, Delamanid and Bedaquiline-Containing Short Regimen For The Treatment Of Rifampicin-Resistant Pulmonary Tuberculosis
Brief Title: Innovating Shorter, All- Oral, Precised, Individualized Treatment Regimen for Rifampicin Resistant Tuberculosis：Contezolid, Delamanid and Bedaquiline Cohort
Acronym: INSPIRE-CODA
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Chest Hospital (Other)
Collaborators: National Medical Center for Infectious Diseases (Unknown)
Responsible Party: Principal Investigator, Chu naihui, Professor, Beijing Chest Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BJCH-202301
Record Dates: First submitted 2023-09-27; First posted 2023-10-13 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Pulmonary Tuberculosis; Rifampicin-resistant Tuberculosis
Keywords: tuberculosis; Rifampicin-resistant; short regimen; contezolid; delamanid
MeSH Terms: conditions — Tuberculosis, Pulmonary; Tuberculosis | interventions — bedaquiline; OPC-67683; contezolid; Levofloxacin; Moxifloxacin; Clofazimine; Linezolid; Cycloserine; Prothionamide; Pyrazinamide; Aminosalicylic Acid; Ethambutol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Short-Term Regimen (Experimental): Intervention will be determined based on Fluoroquinolones(FQs) resistance.
  * For those sensitive to FQs: BDQ DLM CZD LFX(MFX) for 6 months
  * For those resistant to FQs: BDQ DLM CZD CFZ for 6 months
  Interventions: Drug: Bedaquiline; Drug: Delamanid; Drug: Contezolid; Drug: Levofloxacin; Drug: Moxifloxacin; Drug: Clofazimine
- Standard Regimen (Active Comparator): Intervention will be determined based on Fluoroquinolones(FQs) resistance.
  * For those sensitive to FQs: BDQ LZD LFX(MFX) CS CFZ regimen for 6 months, then LFX(MFX) CS CFZ for 12 months
  * For those resistant to FQs: LFX(MFX) will be replaced by Pto, PZA, PAS or EMB
  Interventions: Drug: Bedaquiline; Drug: Levofloxacin; Drug: Moxifloxacin; Drug: Clofazimine; Drug: Linezolid; Drug: Cycloserine; Drug: Prothionamide; Drug: Pyrazinamide; Drug: Para-Aminosalicylic Acid; Drug: Ethambutol

INTERVENTIONS:
Drug: Bedaquiline — Oral, 400mg qd for 2 weeks, then 200 mg 3 times per week
  Other Names: BDQ
Drug: Delamanid — Oral, 100mg bid
  Other Names: DLM
  Arms: Short-Term Regimen
Drug: Contezolid — Oral, 800mg bid
  Other Names: CZD
  Arms: Short-Term Regimen
Drug: Levofloxacin — Oral, 400mg qd for weight <50kg, 600-750mg qd for weight ≥50kg
  Other Names: LFX
Drug: Moxifloxacin — Oral, 400mg qd
  Other Names: MFX
Drug: Clofazimine — Oral, 100mg qd
  Other Names: CFZ
Drug: Linezolid — Oral, 600mg qd
  Other Names: LZD
  Arms: Standard Regimen
Drug: Cycloserine — Oral, 250mg bid
  Other Names: CS
  Arms: Standard Regimen
Drug: Prothionamide — Oral, 600mg qd for weight <50kg, 600-800mg qd for weight ≥50kg
  Other Names: Pto
  Arms: Standard Regimen
Drug: Pyrazinamide — Oral, 1500mg qd for weight <50kg, 1750mg qd for weight ≥50kg
  Other Names: PZA
  Arms: Standard Regimen
Drug: Para-Aminosalicylic Acid — 8000mg qd for weight <50kg, 10000mg qd for weight ≥50kg
  Other Names: PAS
  Arms: Standard Regimen
Drug: Ethambutol — 750mg qd for weight <50kg, 1000mg qd for weight ≥50kg
  Other Names: EMB
  Arms: Standard Regimen

SUMMARY:
The goal of this clinical trial is to compare the efficacy and safety of a Contezolid and Delamanid-Containing short regimen to standard longer regimen in Rifampicin-resistant pulmonary tuberculosis (RR-TB). The main questions it aims to answer are:

* Is the efficacy of short regimen non-inferior to standard regimen?
* Is the short regimen safe enough to replace the standard regimen?

Participants will:

* Be given with either short or standard regimen for RR-TB treatment
* Be asked to complete the scheduled visit as planned.

ELIGIBILITY:
Inclusion criteria:

1. Age ≥18y and <70y when signing informed consent;
2. Initial or re-treatment for pulmonary tuberculosis with:

1) MTB positive in sputum or bronchoalveolar lavage fluid culture at or within 3 months before screening, or MTB positive in molecular test at or within 3 months before screening, and; 2) recorded Rifampicin-resistance at or before screening; 3. Imaging (Chest X-ray or CT scan) proved pulmonary tuberculosis within 1 year before screening; 4. Never used BDQ, DLM or CZD, or the accumulative duration of any of the treatment is not more than 2 weeks 5. For women in childbearing age, negative in pregnancy test and effective contraceptive measures throughout study is required; 6. For men, effective contraceptive measures is required; 7. Willing to participate the study and sign informed consent.

Exclusion criteria:

1. The participant will be excluded by investigator based on the medical history or concomitant diseases such as serious metabolic disease, cardiovascular disease, hepatobiliary disease, renal disease, autoimmune disease, neuropsychiatric disorders, hematological disease, malignant neoplastic disease and so on; or the study will have negative impact on the well-being of the participant, or the participant is considered unable to complete the evaluation by investigator;
2. History of alcohol or drug abuse that the study is considered have negative impact on the well-being of the participant by investigator;
3. HIV positive;
4. Chronic hepatitis with HBsAg, HBeAg and anti-HBC antibody positive, or HBV-DNA>1000 CPs/mL with rising ALT/AST;
5. Allergic to or known hypersensitive to any of study drugs;
6. Extensive (or advanced) pulmonary TB disease: presence of bilateral cavitary disease or extensive parenchymal damage on chest radiography;
7. Hematogenous disseminated pulmonary tuberculosis and serious extrapulmonary tuberculosis (such as tuberculosis in digestive system, urogenital system, osteoarticular tuberculosis, tuberculous meningitis);
8. With any of following risk factors for cardiovascular disease: 1) history of arrhythmia and on consequential treatment; 2) QTcF>500ms on ECG; 3) history of ventricular arrhythmia; 4) torsade de pointe with heart failure, hypokalemia or familial long Q-T syndrome; 5) other possible risk factor for arrythmia;
9. Previous or current optic nerve disorder that may progress or deteriorate during the study by investigator's consideration;
10. Was enrolled within 2 months before screening, or currently in other studies; except for those who participating observational study or in the post-treatment period;
11. Being considered unlikely to survive for more than 6 months by investigator;
12. BMI < 17kg/m2
13. May need surgical procedures based on the evaluation of pulmonary lesions;
14. May continuous use prohibited concomitant medications that is considered not suitable for the study by investigator;
15. Positive in pregnancy test or known pregnancy, breastfeeding, or plan to become pregnant during or within 6 months after the study treatment;
16. Abnormal laboratory test results: 1) Plasma potassium lower than lower limit of normal (LLN); 2) Hb < 8.0 g/dL； 3) platelet count <75,000/mm3； 4) WBC count<3000/mm3； 5）AST/ALT >3×ULN； 6）creatinine>2×ULN；7）total bilirubin>2×ULN, or >1.5×ULN，with abnormal AST or ALT; 8) Albumin < 30g/L

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2023-12-22 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Favourable outcome rate at 24 months after randomization | from randomization to 24 months after
  The proportion of participants with a favourable outcome. A participant's outcome will be classified as favourable if their last two sputum culture results are negative unless they have previously been classified as unfavourable. These two cultures must be taken on separate visits (with ≥28d interval); the latest of which not being earlier than month 23 from randomization.

SECONDARY OUTCOMES:
Unfavourable outcome rate at 24 months after randomization | from randomization to 24 months after
  Including
  1. Death;
  2. Treatment failure
  3. Lost-to-follow-up
  4. Treatment Discontinuation
  5. Ttreatment prolonging
  6. Still on treatment at the end of follow up
  7. Recurrence
Time to culture conversion | from randomization to 24 months after
  Time from treatment initiation to first negative result in sputum culture confirmed by two consecutive cultures with an interval of ≥28d
Grade 3 or higher adverse event rate | from randomization to 24 months after
  Proportion of participants experiencing at least one grade 3 or higher adverse event, or serious adverse event defined by the Division of AIDS severity criteria for adverse events

OTHER OUTCOMES:
Contezolid plasma concentration | 7d±3d after the first dose of contezolid
  To build the population PK model of contezolid with steady-state plasma concentration, measured by blood samples taken at four time points around one administration: ≤15min before and 1h±15min, 2h±15min, 3h±15min after. The index adiministration should be in 7d±3d after the first dose of contezolid.

CONTACTS AND LOCATIONS:
Locations (39):
- China (39):
  - Beijing Chest Hospital affiliated to Capital Medical University, Beijing, Beijing Municipality
  - Changsha Central Hospital, Changsha, China
  - Anhui Chest Hospital, Hefei, China
  - Jiamusi Tumor Hospital, Jiamusi, China
  - Shandong public health clinical center, Shandong, China
  - Xi'an Chest Hospital, Xi'an, China
  - The First Affiliated Hospital of Xinxiang Medical University, Xinxiang, China
  - Hebei Chest Hospital, Shijiazhuang, Hebei
  - Harbin Chest Hospital, Harbin, Heilongjiang
  - Infectious Disease Hospital of Hulunbuir, Hulunbuir, Inner Mongolia
  - Qingdao Chest Hospital, Qingdao, Shandong
  - Taiyuan Fourth People's Hospital, Taiyuan, Shanxi
  - The 8th Medical Center of Chinese Pla General Hospital, Beijing
  - Hunan Province Chest Hospital, Changsha
  - Chongqing Public Heath Treatment Center, Chongqing
  - Dalian Public Health Center, Dalian
  - Fuzhou Pulmonary Hospital of Fujian, Fuzhou
  - Guangzhou Chest Hospital, Guangzhou
  - Heilongjiang Province center for tuberculosis Control and Prevention, Haerbin
  - Second Affiliated Hospital of Hainan Medical University, Haikou
  - Hangzhou Red Cross Hospital, Hangzhou
  - Second People's Hospital of Hohhot, Hohhot
  - Jiamusi Infectious Disease Hospital, Jiamusi
  - Jilin Tuberculosis Hospital, Jilin
  - People's Hospital of Linyi, Linyi
  - Second Hospital of Nanjing, Nanjing
  - Fourth People's Hospital of Nanning, Nanning
  - Guangxi Chest Hospital, Nanning
  - National Medical Center for Infectious Disease, Shanghai
  - Affiliated Hospital of Shaoxing University, Shaoxing
  - Shenyang Chest Hospital, Shenyang
  - Shijiazhuang Fifth Hospital, Shijiazhuang
  - Tianjin Haihe Hospital, Tianjin
  - The 8th Affiliated Hospital of Xinjiang Medical University, Ürümqi
  - Second People's Hospital of Weifang, Weifang
  - Wuhan Institute For Tuberculosis Control, Wuhan
  - First Affiliated Hospital of Xiamen Medical University, Xiamen
  - Henan Provincial Chest Hospital, Zhengzhou
  - Affiliated Hospital of Zunyi Medical University, Zunyi